CLINICAL TRIAL: NCT03080116
Title: Neoadjuvant Degarelix +/- Apalutamide (ARN-509) Followed by Radical Prostatectomy for Intermediate and High-risk Prostate Cancer: a Randomized, Placebo-controlled Trial
Brief Title: Neoadjuvant Degarelix With or Without Apalutamide (ARN-509) Followed by Radical Prostatectomy
Acronym: ARNEO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S58827; 2016-002854-19 (EudraCT Number)
Record Dates: First submitted 2017-02-14; First posted 2017-03-15 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Neoadjuvant Therapy; Androgen Antagonists; Prostatectomy
Keywords: Randomized; Placebo-controlled; Neoadjuvant; Androgen deprivation; Antiandrogen; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARN-509 + degarelix (Experimental): Treatment period of 12 weeks before RP + PLND.
  Interventions: Drug: ARN-509; Drug: Degarelix
- placebo + degarelix (Active Comparator): Treatment period of 12 weeks before RP + PLND.
  Interventions: Drug: Degarelix; Other: Placebo

INTERVENTIONS:
Drug: ARN-509 — 240mg/day (4x60mg tablets, Oral administration: OS)
  Other Names: apalutamide
  Arms: ARN-509 + degarelix
Drug: Degarelix — 1st injection: 120mg Subcutaneous administration (SC) x2, 2nd-3rd SC injection 80mg monthly
Other: Placebo — 4 tablets, per OS
  Arms: placebo + degarelix

SUMMARY:
RATIONALE: Neoadjuvant hormonal therapy using luteinizing hormone releasing hormone (LHRH) agonists and/or anti-androgens has already demonstrated to downstage primary prostate cancer in patients treated by radical prostatectomy without a survival benefit. There is no evidence yet of a survival impact of LHRH antagonist (LHRHa) +/- new-generation anti-androgens in this setting. Thus novel studies are needed to assess this treatment combination.

PURPOSE: To assess the difference in treatment antitumor effect between arms by measuring pathological tumor volume with minimal residual disease (MRD) following radical prostatectomy + pelvic lymph-node dissection (RP + PLND) for intermediate or high-risk prostate cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: To assess the difference in antitumor effect between the treatment arms by measuring MRD following radical prostatectomy.

SECONDARY OBJECTIVES: To measure differences between study arms in

* Proportions of post neoadjuvant prostate specific antigen (PSA) ≤ 0.3 ng/ml as a predictor of prostate cancer mortality
* T down-staging, complete pathological response, PSA kinetics, Testosterone kinetics, operation time, blood loss, grade of surgical difficulty
* New generation hybrid imaging 68Ga PSMA (Prostate-Specific Membrane Antigen) PET/MR (Positron emission tomography/Magnetic Resonance) derived parameters
* Early biochemical recurrence as prognostic factor of prostate cancer mortality
* Transcriptome and genome
* Tissue microarrays (TMA) protein expression (DNA repair, resistance etc.) by immunohistochemistry
* Perioperative safety and tolerability
* Quality of life, erection recovery, continence through validated preoperative and postoperative questionnaires pre and postop (IEEF5, ICIQ, EORTC QLQ-C30)

OUTLINE: interventional, single center, phase II, randomized, double blind, placebo controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
2. Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations
3. Male aged 18 years or older (within 80 years)
4. Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
5. Diagnosis of intermediate (at least 2 of the following factors: cT2b, biopsy GS 7, PSA 10-20ng/ml) or high-risk prostatic adenocarcinoma (clinical stage≥T2c and/or biopsy GS≥8 and/or PSA>20ng/ml), cN0-cN1, cM0.
6. Patient amenable for open or robotic radical prostatectomy + pelvic lymph node dissection
7. ECOG performance status: 0-1
8. Adequate organ function as defined by the following criteria:

   * White blood cells (WBC) ≥ 4.0 x109/L
   * Platelet count ≥ 100 x109/L
   * Hemoglobin ≥9 g/dl
   * Creatinine ≤ 2 x ULN
   * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x upper limit of normality (ULN)
   * Total serum bilirubin ≤1.5 x ULN.

Exclusion Criteria:

1. Previous surgical/endoscopic treatments for prostatic disease
2. Herbal and non-herbal products that in the opinion of the investigator may decrease PSA levels
3. cM1 disease
4. Any contraindication for PET or MR investigations
5. History of seizure or condition that may pre-dispose to seizure (e.g., prior stroke within 1 year prior to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy)
6. Medications known to lower the seizure threshold
7. History of:

   * Any prior malignancy (other than adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer currently in complete remission) within 5 years prior to randomization
   * Severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
   * Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic BP ≥100 mmHg). Patients with a history of uncontrolled hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
   * Gastrointestinal disorder affecting absorption
8. Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD) | After 12 weeks of neoadjuvant therapy + RP + PLND
  Proportions of MRD between arms. MRD: tumor volume ≤ 0.25 cm3

SECONDARY OUTCOMES:
Difference in proportions of pathological downstage | After 12 weeks of neoadjuvant therapy + RP + PLND
  Any decrease in T stage from clinical to pathological stage
Complete pathological response rates | After 12 weeks of neoadjuvant therapy + RP + PLND
  Difference in proportions of complete pathological response (no evidence of tumour in the postoperative specimen) between arms.
Difference in proportions of patients with pN1 disease. | After 12 weeks of neoadjuvant therapy + RP + PLND
  Difference in proportions of lymph node invasion between arms
Proteins expression in prostatic tumour TMA's (tissue microarrays) | After 12 weeks of neoadjuvant therapy + RP + PLND
  Intensity of immunoreactivity and percentage of immunoreactive cells for, selected markers between arms. The TMA's will be produced from the formalin-fixed paraffin-embedded (FFPE) specimen of the RP.
Transcriptome analysis by microarray expression platform | At baseline and after 12 weeks of neoadjuvant therapy + RP + PLND
  To assess differences in the transcriptome in tumour tissue on formalin-fixed paraffin-embedded (FFPE) specimens: clinical-grade high-density oligonucleotide microarray expression platform and cloud-based informatics pipeline to interrogate 1.4M probe sets representing all known ~46K genes and non-coding RNAs.
Pathway profiling and Gene Set Enrichment Analyses | At baseline and after 12 weeks of neoadjuvant therapy + RP + PLND
  To assess differences in the transcriptome in tumour tissue on formalin-fixed paraffin-embedded (FFPE) specimens. Pathway profiling and Gene Set Enrichment Analyses will also be used to generate pathway scores for the 'androgen receptor signaling pathway'; determination of pathway scores for the DNA damage checkpoints and the different DNA repair pathways.
Genomic subtyping by exome-sequencing | At baseline and after 12 weeks of neoadjuvant therapy + RP + PLND
  Genomic subtyping (e.g., ERG, SPINK1, SPOP, FOXA1, PTEN, circulating nucleic acids (CNA) data...) will be performed based on exome-sequencing data. The exome and CNA data will be linked with the transcriptome data on androgen regulation and DNA repair pathways.
PSA kinetics | Up to 40 months
  Changes of PSA during time and comparison of PSA values and changes between arms.
Testosterone kinetics | Up to 40 months
  Comparison of total and free serum testosterone and testosterone change between arms
PSA nadir </=0.3ng/ml after neoadjuvant treatment | After 12 weeks of neoadjuvant therapy before RP + PLND
  Differences in proportions of PSA nadir </=0.3ng/ml after neoadjuvant treatment.
  PSA nadir after neoadjuvant therapy and before external beam radiotherapy (EBRT) is an important biomarker of hormonal response and an independent prognostic factor of prostate cancer survival.
Peri-operative features | up to (about) 5 hours
  Differences in peri-operative features (operative time, blood loss, grade of surgical difficulty...) will be collected to evaluate the possible effect of treatment on surgical intervention.
Differences in proportions of surgical complications between arms | Up to 6 weeks post RP + PLND
  Clavien-Dindo classification will be implemented to assess differences in surgical complications between the two arms.
Continence | Up to 40 months
  Assessment of continence rates through validated preoperative and postoperative questionnaire (ICIQ)
Quality of life | Up to 40 months
  Assessment of Quality of life through validated preoperative and postoperative questionnaire (EORTC QLQ-C30)
Erection state | Up to 40 months
  Assessment of erection state through validated preoperative and postoperative questionnaire (IEEF5)
Survival | Up to 36 months
  Three years biochemical recurrence free survival
Standardized Uptake Value (SUV) on pelvic [68]Ga PSMA PET/MR per arm | At baseline and after 12 weeks of neoadjuvant therapy + RP + PLND
  Standardized Uptake Value (SUV) change (delta) per arm comparing SUV values before and after treatment
Standardized Uptake Value (SUV) on pelvic [68]Ga PSMA PET/MR between arms | After 12 weeks of neoadjuvant therapy + RP + PLND
  SUV delta between the two arms.
Standardized Uptake Value (SUV) on pelvic [68]Ga PSMA PET/MR and tumour volume | After 12 weeks of neoadjuvant therapy + RP + PLND
  Correlation between SUV values and the tumour volume (TV) in the RP correspondent volume of interest (VOI) at definitive pathology
Standardized Uptake Value (SUV) on prostate [68]Ga PSMA PET/MR and Immunohistochemistry | After 12 weeks of neoadjuvant therapy + RP + PLND
  Correlation between SUV values and PSMA expression at Immunohistochemistry
Magnetic resonance (MR) and tumor volume (TV) per arm | At baseline and after12 weeks of neoadjuvant therapy + RP + PLND
  Change of magnetic resonance (MR) tumor volume (TV): Tumor volume (TV) change (delta) per arm comparing TV values before and after treatment
Magnetic resonance (MR) and tumor volume (TV) between arms | At baseline and after12 weeks of neoadjuvant therapy + RP + PLND
  Change of magnetic resonance (MR) tumor volume (TV):TV deltas between the two arms.
PI-RADS between arms at MR | After 12 weeks of neoadjuvant therapy + RP + PLND
  Proportion of PI-RADS between arms
PI-RADS score and Gleason score | After 12 weeks of neoadjuvant therapy + RP + PLND
  Correlation between PI-RADS score and pathology Gleason score
Down-staging at imaging | At baseline and after 12 weeks of neoadjuvant therapy + RP + PLND
  Proportion of down-staging
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From patient inclusion until RP + PLND
  Frequencies of adverse events (AE), severe adverse events (SAE) and Suspected Unexpected Serious Adverse Reaction (SUSAR)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joniau, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-brabant, Belgium

REFERENCES:
- [Derived] Tosco L, Laenen A, Gevaert T, Salmon I, Decaestecker C, Davicioni E, Buerki C, Claessens F, Swinnen J, Goffin K, Oyen R, Everaerts W, Moris L, De Meerleer G, Haustermans K, Joniau S; P.E.A.R.L. (ProstatE cAncer Research Leuven). Neoadjuvant degarelix with or without apalutamide followed by radical prostatectomy for intermediate and high-risk prostate cancer: ARNEO, a randomized, double blind, placebo-controlled trial. BMC Cancer. 2018 Apr 2;18(1):354. doi: 10.1186/s12885-018-4275-z. PMID 29606109